CLINICAL TRIAL: NCT01887223
Title: Early Transconjunctival Needling Revision With 5-fluorouracil Versus Medical Treatment in Encapsulated Blebs: a 12-month Prospective Study
Brief Title: Transconjunctival Needling Revision Versus Medical Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ricardo Suzuki, Assistant professor of Ophthalmology at HCFMUSP, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNRVMT-RS
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Encapsulated blebs; trabeculectomy failure; glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Latanoprost; dorzolamide; Brimonidine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transconjunctival needling revision (Experimental): Eyes with primary glaucoma surgery failure with encapsulated bleb submitted to surgical revision
  Interventions: Procedure: Transconjunctival needling revision
- Medical treatment (Active Comparator): Eyes with primary glaucoma surgery failure with encapsulated blebs were treated with medical treatment (hypotensive eye drops)
  Interventions: Drug: Medical treatment

INTERVENTIONS:
Procedure: Transconjunctival needling revision — Surgical revision. A 25 Gauge needle was inserted under the subconjunctival space and perforate the encapsulated bled. The encapsulated bleb was ruptured with sweeping movement up and down, back and forth.
  Arms: Transconjunctival needling revision
Drug: Medical treatment — Hypotensive eye drops are initialized one by one regarding intraocular pressure control. Nonspecific beta blocker and/or prostaglandin, followed by carbonic anhydrase inhibitors and/or selective alpha agonist.
  Other Names: Timoptol 0,5%; Xalatan; Trusopt; Alphagan
  Arms: Medical treatment

SUMMARY:
When the glaucoma filtering surgery failures (intraocular pressure rises again), the options is start to use the hypotensive eye drops again (medical treatment). However, in some cases (encapsulated blebs), there is a simple surgical revision that can revival the primary failure surgery. It calls transconjunctival needling revision. In this study, the investigators compare the efficacy of this revision versus medical treatment in 12-month follow up in eyes with encapsulated blebs.

DETAILED DESCRIPTION:
To compare the efficacy of transconjunctival needling revision (TNR) with 5-fluorouracil versus medical treatment (MT) in glaucomatous eyes with uncontrolled intraocular pressure (IOP) due to encapsulated bleb after trabeculectomy Prospective, randomized, interventional study. A total of forty eyes of 39 patients with elevated IOP and encapsulated bleb diagnosed at maximum 5 months after primary trabeculectomy with mitomycin C were included. The eyes were randomized to either TNR with 5-fluorouracil or MT (hypotensive eyedrops). A maximum of two TNR per patient was allowed in the needling arm. All eyes were followed up for 12 months. Success of treatment was defined as IOP ≤ 18mmHg and 20% reduction from baseline at last follow up.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with encapsulated blebs developed in 5 months or less following primary glaucoma filtering surgery (trabeculectomy) and intraocular pressure >= 20mmHg

Exclusion Criteria:

* Previous other ocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Remo Susanna Jr., MD, Study Chair — University of Sao Paulo General Hospital; Ricardo Suzuki, MD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Costa VP, Correa MM, Kara-Jose N. Needling versus medical treatment in encapsulated blebs. A randomized, prospective study. Ophthalmology. 1997 Aug;104(8):1215-20. doi: 10.1016/s0161-6420(97)30155-9. PMID 9261306
- [Derived] Suzuki R, Susanna R Jr. Early transconjunctival needling revision with 5-fluorouracil versus medical treatment in encapsulated blebs: a 12-month prospective study. Clinics (Sao Paulo). 2013 Oct;68(10):1376-9. doi: 10.6061/clinics/2013(10)14. PMID 24212847